CLINICAL TRIAL: NCT00105560
Title: Phase II Study of Craniospinal and Posterior Fossa Irradiation Using Proton Beam Radiotherapy for Medulloblastoma and Pineoblastoma: Assessment of Acute and Long Term Sequelae
Brief Title: Proton Beam Radiation Therapy in Treating Young Patients Who Have Undergone Biopsy or Surgery for Medulloblastoma or Pineoblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nancy J. Tarbell, M.D., Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415841; P01CA021239 (NIH); MGH-99-271 (Other: Massachusetts General Hospital)
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Brain and Central Nervous System Tumors; Long-term Effects Secondary to Cancer Therapy in Children
Keywords: long-term effects secondary to cancer therapy in children; untreated childhood medulloblastoma; untreated childhood pineoblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation therapy (Experimental): This is a single arm study of radiation therapy with protons to standard doses.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Radiation therapy with proton beam to standard doses

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers radiation directly to the area where a tumor was surgically removed may kill any remaining tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying how well proton beam radiation therapy works in treating young patients who have undergone biopsy or surgery for medulloblastoma or pineoblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 3-year incidence and severity of ototoxicity in young patients with medulloblastoma or pineoblastoma treated with adjuvant proton beam craniospinal and posterior fossa radiotherapy.
* Determine the incidence of primary hypothyroidism and other endocrine dysfunction (neuroendocrine and end organ) in patients treated with this regimen.
* Determine the incidence and severity of neurocognitive abnormalities in patients treated with this regimen.
* Determine the acute side effects of this regimen, including esophagitis, upper and lower gastrointestinal tract disease, and weight loss, in these patients.
* Determine the 3-year progression-free survival rate of patients treated with this regimen.

OUTLINE: Patients are stratified according to risk (standard vs high).

Patients receive proton beam craniospinal and posterior fossa radiotherapy once daily 5 days a week for 6-8 weeks*.

NOTE: *Unless otherwise specified by a co-existing protocol.

Patients undergo neurocognitive evaluation at baseline or within 3 months after completion of radiotherapy and then at 1, 3, and 5 years. Patients also undergo endocrine evaluation at baseline and then annually for 5 years; and audiology evaluation at baseline, before each course of cisplatin-based chemotherapy (if receiving this), and then annually for 5 years.

After completion of study treatment, patients are followed every 3-6 months for 2-5 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed medulloblastoma or pineoblastoma

  * Standard-risk or high-risk disease
* Must have undergone biopsy or attempted surgical resection of the tumor within the past 35 days
* Requires craniospinal irradiation

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 1 prior chemotherapy regimen
* No prior IV or intrathecal methotrexate
* No prior intrathecal thiotepa
* Concurrent cisplatin-based chemotherapy, including chemotherapy administered on another study, allowed

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Tarbell, MD, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yock TI, Yeap BY, Ebb DH, Weyman E, Eaton BR, Sherry NA, Jones RM, MacDonald SM, Pulsifer MB, Lavally B, Abrams AN, Huang MS, Marcus KJ, Tarbell NJ. Long-term toxic effects of proton radiotherapy for paediatric medulloblastoma: a phase 2 single-arm study. Lancet Oncol. 2016 Mar;17(3):287-298. doi: 10.1016/S1470-2045(15)00167-9. Epub 2016 Jan 30. PMID 26830377
- [Derived] Vatner RE, Niemierko A, Misra M, Weyman EA, Goebel CP, Ebb DH, Jones RM, Huang MS, Mahajan A, Grosshans DR, Paulino AC, Stanley T, MacDonald SM, Tarbell NJ, Yock TI. Endocrine Deficiency As a Function of Radiation Dose to the Hypothalamus and Pituitary in Pediatric and Young Adult Patients With Brain Tumors. J Clin Oncol. 2018 Oct 1;36(28):2854-2862. doi: 10.1200/JCO.2018.78.1492. Epub 2018 Aug 17. PMID 30118397

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 59
Completed | 58
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.6 [5.1 to 9.9]
Age, Customized [Count of Participants; unit: Participants]
  < 8 Years | 37
  ≥ 8 Years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59
Histological Subtype (Dominant Pattern) [Count of Participants; unit: Participants]
  Classic | 45
  Desmoplastic or Nodular Variant | 6
  Anaplastic or Large Cell Variant | 8
Risk Group [Count of Participants; unit: Participants] — Intermediate risk is defined as M0 patients with <1·5 cm² of residual disease but with anaplastic or large cell variant. If residual disease at the primary site was greater than or equal to 1·5 cm² on axial MRI, then they would be classified as high risk if they had no other evidence of metastatic disease.
  Participants
    Standard | 39
    Intermediate | 6
    High | 14
Posterior Fossa Syndrome [Count of Participants; unit: Participants]
  Yes | 14
  No | 45
Ventriculoperitoneal Shunt [Count of Participants; unit: Participants]
  Yes | 12
  No | 47
Enrolled on a Children's Oncology Group Protocol [Number; unit: participants] — The alphanumeric codes next to the 'yes' represent Children's Oncology Group protocol numbers
  participants
    Yes : ACNS0331 | 8
    Yes : ACNS0332 | 2
    Yes : ACNS0334 | 1
    Yes : A9961 | 1
    No | 47
Boost Field [Count of Participants; unit: Participants]
  Tumor Bed Involved Field | 36
  Posterior Fossa | 23
Boost Dose [Count of Participants; unit: Participants] — Dose measured as Gray (Gy) Relative Biological Effectiveness (RBE)
  Participants
    54 GyRBE | 57
    >54 GyRBE | 2
Craniospinal Radiation Doses [Count of Participants; unit: Participants]
  18-27 GyRBE | 45
  36 GyRBE | 14
Hypothalamus Mean Dose (D50) [Count of Participants; unit: Participants] — D50 (the half maximal inhibitory dose) is the dose of radiation that is required for 50% inactivation of a tumor cell population.
  Participants
    <40 GyRBE | 37
    ≥40 GyRBE | 22
Cochlear Mean Dose to Each Ear (D50) [Number; unit: Ears]
  <30 GyRBE | 61
  ≥30 GyRBE | 57
Cisplatin Cumulative Dose [Number; unit: participants] — Cisplatin cumulative dose information is not available for eight of the participants
  participants
    ≤300 mg/m2 | 17
    >300 mg/m2 | 34
Use of Photons for <20% radiation dose [Count of Participants; unit: Participants]
  Yes | 6
  No | 53

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Ototoxicity
Description: Percentage participants who experienced ototoxicity as measured by Common Toxicity Criteria for Adverse Events (CTCAE) v3.0 after the completion of radiation therapy in the overall participant population and by baseline measure subgroups. Incidence is shown after follow-up of 3 years, 5 years, 7 years, and 10 years.
Time Frame: 3 Years, 5 years, 7 years, 10 years
Population: The overall study population after the stated durations of follow-up. Follow-up is ongoing and data is not yet available for the 10 year time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Radiation Therapy - 3 Years Follow-up; Radiation Therapy - 5 Years Follow-up; Radiation Therapy - 7 Years Follow-up: radiation therapy: Radiation therapy with proton beam to standard doses
Arm/Group | Radiation Therapy - 3 Years Follow-up | Radiation Therapy - 5 Years Follow-up | Radiation Therapy - 7 Years Follow-up
Number analyzed (Participants) | 59 | 59 | 59
percentage of participants
  All Participants | 12 [4 to 25] | 16 [6 to 29] | 16 [6 to 29]
  Standard Risk: number analyzed (Participants) | 39 | 39 | 39
  Standard Risk | 15 [4 to 31] | 20 [7 to 38] | 20 [7 to 38]
  Intermediate-high risk: number analyzed (Participants) | 20 | 20 | 20
  Intermediate-high risk | 7 [0 to 29] | 7 [0 to 29] | 7 [0 to 29]
  Male: number analyzed (Participants) | 33 | 33 | 33
  Male | 4 [0 to 19] | 4 [0 to 19] | 4 [0 to 19]
  Female: number analyzed (Participants) | 26 | 26 | 26
  Female | 20 [6 to 40] | 27 [9 to 49] | 27 [9 to 49]
  <8 years old: number analyzed (Participants) | 37 | 37 | 37
  <8 years old | 15 [5 to 32] | 20 [7 to 38] | 20 [7 to 38]
  ≥8 years old: number analyzed (Participants) | 22 | 22 | 22
  ≥8 years old | 6 [0 to 25] | 6 [0 to 25] | 6 [0 to 25]
  Vetriculoperitoneal shunt: number analyzed (Participants) | 12 | 12 | 12
  Vetriculoperitoneal shunt | 22 [3 to 53] | 22 [3 to 53] | 22 [3 to 53]
  No vetriculoperitoneal shunt: number analyzed (Participants) | 47 | 47 | 47
  No vetriculoperitoneal shunt | 10 [2 to 24] | 14 [4 to 29] | 14 [4 to 29]
  Cisplatin total dose ≤300 mg/m2: number analyzed (Participants) | 17 | 17 | 17
  Cisplatin total dose ≤300 mg/m2 | 18 [2 to 46] | 18 [2 to 46] | 18 [2 to 46]
  Cisplatin total dose >300 mg/m2: number analyzed (Participants) | 34 | 34 | 34
  Cisplatin total dose >300 mg/m2 | 12 [3 to 28] | 17 [5 to 35] | 17 [5 to 35]

2. Secondary Outcome: Cumulative Incidence of Endocrine Dysfunction (Neuroendocrine and End Organ Defects) at 3 Years
Description: Percentage of participants who experienced endocrine dysfunction (neuroendocrine and end organ defects) after 3 years of follow-up (as determined by CTCAE 3.0). Incidence is grouped by hormone type and risk group
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Radiation Therapy - Overall Study Population; Radiation Therapy - Standard Risk Group; Radiation Therapy Intermediate-High Risk: radiation therapy: Radiation therapy with proton beam to standard doses
Arm/Group | Radiation Therapy - Overall Study Population | Radiation Therapy - Standard Risk Group | Radiation Therapy Intermediate-High Risk
Number analyzed (Participants) | 59 | 39 | 20
percentage of participants
  Any hormone deficit | 27 [16 to 39] | 28 [15 to 43] | 25 [9 to 46]
  Growth hormone deficit | 22 [12 to 33] | 23 [11 to 37] | 20 [6 to 40]
  Thyroid deficiency | 12 [5 to 22] | 10 [3 to 22] | 15 [4 to 34]
  Adrenal or cortisol deficit | 5 [1 to 13] | 3 [0 to 12] | 10 [2 to 28]
  Sex hormone deficit | 3 [1 to 11] | 3 [0 to 12] | 5 [0 to 21]

3. Secondary Outcome: Cumulative Incidence of Endocrine Dysfunction (Neuroendocrine and End Organ Defects) at 5 Years
Description: Percentage of participants who experienced endocrine dysfunction (neuroendocrine and end organ defects) after 5 years of follow-up (as determined by CTCAE 3.0). Incidence is shown by hormone type and risk group.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Radiation Therapy - Intermediate-High Risk: radiation therapy: Radiation therapy with proton beam to standard doses
Arm/Group | Radiation Therapy - Overall Study Population | Radiation Therapy - Standard Risk Group | Radiation Therapy - Intermediate-High Risk
Number analyzed (Participants) | 59 | 39 | 20
percentage of participants
  Any hormone deficit | 55 [41 to 67] | 58 [40 to 72] | 50 [26 to 70]
  Growth hormone deficit | 46 [33 to 59] | 50 [33 to 65] | 40 [18 to 61]
  Thyroid deficiency | 21 [11 to 32] | 21 [10 to 35] | 20 [6 to 40]
  Adrenal or cortisol deficit | 9 [3 to 17] | 3 [0 to 12] | 20 [6 to 40]
  Sex hormone deficit : Overall study population | 3 [1 to 11] | 3 [0 to 12] | 5 [0 to 21]

4. Secondary Outcome: Cumulative Incidence of Endocrine Dysfunction (Neuroendocrine and End Organ Defects) at 7 Years
Description: Percentage of participants who experienced endocrine dysfunction (neuroendocrine and end organ defects) after 7 years of follow-up, as determined by CTCAE 3.0. Incidence is shown by hormone type and risk group
Time Frame: 7 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy - Overall Study Population | Radiation Therapy - Standard Risk Group | Radiation Therapy - Intermediate-High Risk
Number analyzed (Participants) | 59 | 39 | 20
percentage of participants
  Any hormone deficit | 63 [48 to 75] | 68 [49 to 82] | 50 [26 to 70]
  Growth hormone deficit | 55 [40 to 68] | 62 [42 to 76] | 40 [18 to 61]
  Thyroid deficiency | 26 [15 to 38] | 25 [12 to 40] | 29 [9 to 53]
  Adrenal or cortisol deficit | 9 [3 to 17] | 3 [0 to 12] | 20 [6 to 40]
  Sex hormone deficit : Overall study population | 3 [1 to 11] | 3 [0 to 12] | 5 [0 to 21]

5. Secondary Outcome: Cumulative Incidence of Endocrine Dysfunction (Neuroendocrine and End Organ Defects) at 7 Years
Description: percentage of participants who experienced endocrine dysfunction (neuroendocrine and end organ defects) as determined by CTCAE 3.0) at year 3, year 5, and year 7 of follow-up.
Time Frame: 3 years, 5 years, 7 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy - 3 Years Follow-up | Radiation Therapy - 5 Years Follow-up | Radiation Therapy - 7 Years Follow-up
Number analyzed (Participants) | 59 | 59 | 59
percentage of participants
  Any hormone deficit | 27 [16 to 39] | 55 [41 to 67] | 63 [48 to 75]
  Growth hormone deficit | 22 [12 to 33] | 46 [33 to 59] | 55 [40 to 68]
  Thyroid deficiency | 12 [5 to 22] | 21 [11 to 32] | 26 [15 to 38]
  Adrenal or cortisol deficit | 5 [1 to 13] | 9 [3 to 17] | 9 [3 to 17]
  Sex hormone deficit | 3 [1 to 11] | 3 [1 to 11] | 3 [1 to 11]

6. Secondary Outcome: Mean Change Per-Year in Neurocognitive Outcomes
Description: The mean change per-year in neurocognitive outcomes as assessed by Wechsler Intelligence Scale for Children version 4 (WISC-IV). The test measures the Full Scale Intelligence Quotient (FSIQ) of children with the use of four indices; the Verbal Comprehension Index (VCI), Perceptual Reasoning Index (PRI), working memory test, and a processing speed test. FSIQ and the four indices are all assessed on a bell curve scale that has an average score of 100 and standard deviation of 15 points in the general population, meaning on average 68% of test takers would be within +/- 15 points of 100 and 95% within +/- 30 points. Higher scores represent higher intelligence and lower score represent reduced intelligence. Participants were assessed for changes in score with the use of repeated testing during a median follow-up time of 5.2 years. Repeated measures were taken at baseline, 1, 3, 5, and 7 years or until the participant was not available for evaluation (whichever comes first).
Time Frame: Baseline, 1, 3, 5, 7 years
Population: The study participants that were evaluated for changes in neurocognitive outcomes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 54
units on a scale
  FSIQ | -1.5 [-2.1 to -0.9]
  VCI: number analyzed (Participants) | 53
  VCI | -1.3 [-2.0 to -0.7]
  PRI: number analyzed (Participants) | 53
  PRI | -.4 [-1.0 to 0.3]
  Working Memory: number analyzed (Participants) | 41
  Working Memory | -0.8 [-1.8 to 0.3]
  Processing speed: number analyzed (Participants) | 49
  Processing speed | -2.4 [-3.2 to -1.6]

7. Secondary Outcome: Progression Free Survival
Description: The percentage of participants with progression free survival after five, seven, and ten years in the overall population and by risk and histological group.
Time Frame: 5 years, 7 years, 10 years
Population: Follow-up is ongoing and data is not yet available for the 10 year follow-up time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants surviving
Arm/Group | Radiation Therapy - 5 Years Follow-up | Radiation Therapy - 7 Years Follow-up
Number analyzed (Participants) | 59 | 59
percentage of participants surviving
  All Participants | 80 [67 to 88] | 75 [61 to 84]
  Standard Risk | 85 [69 to 93] | 81 [64 to 91]
  Intermediate-high risk | 70 [45 to 85] | 63 [37 to 81]
  Classic or desmoplastic histological subtype | 80 [67 to 89] | 75 [61 to 85]
  Anaplastic or large cell histological subtype | 75 [31 to 93] | 75 [31 to 93]

8. Secondary Outcome: Overall Survival
Description: the percentage of participants surviving after five and seven years and at the end of follow-up in the overall population. Survival is shown by risk and histological group.
Time Frame: 5 years, 7 years, 10 years
Population: Follow-up for the 10 year follow-up is still ongoing and the data is not yet available.
Measure: Number (95% Confidence Interval); unit: percentage of participants surviving
Arm/Group | Radiation Therapy - 5 Years Follow-up | Radiation Therapy - 7 Years Follow-up
Number analyzed (Participants) | 59 | 59
percentage of participants surviving
  All Participants | 83 [70 to 90] | 81 [67 to 89]
  Standard Risk | 86 [70 to 94] | 86 [70 to 94]
  Intermediate-high risk | 75 [50 to 89] | 68 [42 to 84]
  Classic or desmoplastic histological subtype | 84 [70 to 92] | 82 [67 to 90]
  Anaplastic or large cell histological subtype | 75 [31 to 93] | 75 [31 to 93]

ADVERSE EVENTS:
Time Frame: Through study completion, median duration of 7 years
Description: Acute toxicity is assessed weekly during craniospinal irradiation (CSI) treatment and late side effects/complications are assessed during routine clinic visits starting at 90 days after the completion of radiation therapy. Participants were assessed for toxicity for the duration of followup, meaning until the patient withdraws from the study, is taken off the protocol, or dies.
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 13/59
Serious Adverse Events (participants affected / at risk) | 13/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy (N=59)
Neutropenia (Investigations) | 5
Lymphopenia (Investigations) | 7
Stroke (Nervous system disorders) | 1
esophhagitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy (N=59)
Alopecia (Skin and subcutaneous tissue disorders) | 59
Fatigue (General disorders) | 45
Anorexia (Metabolism and nutrition disorders) | 35
Nausea (Gastrointestinal disorders) | 34
Vomiting (Gastrointestinal disorders) | 32
Radiation dermatitis (scalp or back) (Skin and subcutaneous tissue disorders) | 21
Headache (Nervous system disorders) | 17
Weight Loss (Investigations) | 10
Neutropenia (Blood and lymphatic system disorders) | 42
Lymphopenia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Cataracts (Eye disorders) | 16
Obesity (Metabolism and nutrition disorders) | 7
CNS brainstem injury (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 28
Depression (Psychiatric disorders) | 4
Scoliosis (Musculoskeletal and connective tissue disorders) | 5
Truncal muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Nystagmus (Nervous system disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes